CLINICAL TRIAL: NCT05476718
Title: The Effect of Kinesio Taping on Pain and Functionality in the Rehabilitation Process After Lumbar Disc Surgery
Brief Title: Kinesio Taping in Patients After Lumbar Disc Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gulsah, Master student, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Gülşah
Record Dates: First submitted 2022-06-29; First posted 2022-07-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Lumbar Disc Surgery; Post Operative Pain
Keywords: Lumbar Disc Surgery; Post Operative Pain; Functionality; Rehabilitation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: In this study, which was designed as a randomized controlled study (pretest-posttest control group design), Kinesio and placebo groups were formed as the experimental and control groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: In a randomized, placebo-controlled experimental trial, the participants and data analyzer will be blinded, and the researcher will be blinded to group assignments. Randomizer org site will be used for random assignment of groups as Kinesio or placebo (httpp://www.random.org/lists/). Index cards prepared by simple randomization by the researcher who did not participate in the clinical part of the study will be placed in closed opaque envelopes and sequence numbers will be written on the envelopes. Envelopes will be retained by the clinical secretary who did not participate in the study. The research data will be entered into the computer database by the researcher as coded as A and B, statistical analyzes will be carried out by the researcher who did not participate in the data collection phase according to this code, and the research report will be written in coded form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesio group (Active Comparator): The tape will be applied in the first 24 hours postoperatively and on the 5th, 10th, 15th days of the surgery. The posterior superior iliac spine (PSI) and 12th thoracic vertebra (T12) will be marked while the participant is sitting in a comfortable position. Tape application will be made bilaterally between PSI and T12 with tapes cut in an "I" shape along the erector spine muscles. The anchor and end parts of the tape will be rounded. The anchor part will be glued without tension. Afterward, individuals are asked to flex and rotate their trunks as much as possible, and the middle part of the band is slightly stretched 10-15%; After the spine is brought to its normal anatomical position, the tip will be glued without tension. After sticking, the tape will be manually activated. This transaction will be carried out by both parties. After the tape adheres, individuals will be asked to keep the tape for five days until the next taping.
  Interventions: Other: Kinesio taping
- placebo group (Placebo Comparator): The tape will be applied in the first 24 hours postoperatively and on the 5th, 10th, 15th days of the surgery. The placebo-tape application will be applied the lumbar region in a tension-free and horizontal form, while the spine is in a neutral position without positioning the patients. After sticking, the tape will be manually activated. After the tape adheres, individuals will be asked to hold the tape for five days until the next taping.
  Interventions: Other: placebo taping

INTERVENTIONS:
Other: Kinesio taping — Patients will be informed about the study on the first day of their hospitalization and the Introductory Information Form, Visual Analogue Scale, and Oswestry Disability Index will be filled in by the patients. 24 hours after the operation, 20 minutes of training will be given to the patient and their relatives on the use of a pedometer and home care, and the first tape will be applied. After discharge, the renewal of the bands will be carried out on the postoperative 1th- 5th-10th-15th days when the patients come to the hospital for post-op evaluation. The clinical recovery of the operation area will be done by the investigative physician. In the follow-ups, evaluations will be made with the Visual Analog Scale, Medication Tracking Form, Oswestry Disability Index,Functional Low Back Pain Scale, Kinesio Tracking Form, and Gait Tracking Form.
  Arms: kinesio group
Other: placebo taping — Patients will be informed about the study on the first day of their hospitalization and the Introductory Information Form, Visual Analogue Scale, and Oswestry Disability Index will be filled in by the patients. 24 hours after the operation, 20 minutes of training will be given to the patient and their relatives on the use of a pedometer and home care, and the first tape will be applied. After discharge, the renewal of the bands will be carried out on the postoperative 1th-5th-10th-15th days when the patients come to the hospital for post-op evaluation. The clinical recovery of the operation area will be done by the investigative physician. In the follow-ups, evaluations will be made with the Visual Analog Scale, Medication Tracking Form, Oswestry Disability Index,Functional Low Back Pain Scale, Kinesio Tracking Form, and Gait Tracking Form.
  Arms: placebo group

SUMMARY:
In this study, it will be determined whether Kinesio-tape is an effective and reliable application in reducing pain and maintaining functionality after lumbar disc surgery, and its effect on the rehabilitation process will be evaluated.

DETAILED DESCRIPTION:
According to the 2019 Global Burden of Disease Survey published by the World Health Organization, the problems that contribute most to disability at the global level are musculoskeletal problems. Approximately 1.71 billion people in the world have musculoskeletal diseases (MSD), and low back pain is among the leading causes of disability in 160 countries. According to Turkey's 2019 Global Burden of Disease results, low back pain ranks first among the top ten causes of life years lost due to disability.

Low back pain is also the most common symptom of lumbar disc herniation. Pharmacological, non-pharmacological, and surgical treatment methods can be applied according to the nature of the damage in lumbar disc herniation. Mild to moderate back and leg pain, disability, limitation of function, and decrease in work performance are among the most common problems encountered by patients after surgical intervention for lumbar disc herniation. It is important to reduce low back pain and increase functionality after surgery. Numerous treatments have been researched for low back pain. Kinesio-tape application is gaining popularity around the world and has recently been seen as a preferred option for low back pain.

Kinesio-tape is a rehabilitation technique, designed to facilitate the natural healing process after trauma/inflammation by providing stability and support to muscles and joints. In recent years, its use has been increasing in musculoskeletal problems, neurological, rheumatic, vascular, and lymphatic problems. The Kinesio-tape is easy to apply, it can stay on the skin for a week; It is thought that it can be easily used by patients because it does not require constant effort and time, as in other physical therapy methods such as exercise. Although it has been suggested that Kinesio taping can be used together with traditional analgesic methods to reduce low back pain, no research has been found on the use of Kinesio tape after lumbar disc surgery. This study, it was aimed to determine whether Kinesio-taping is an effective and safe application in reducing post-operative lumbar pain and preserving functionality and to evaluate its effect on the rehabilitation process.

The study, planned as a randomized controlled experimental study, will be conducted with 80 patients (40 Kinesio and 40 placebo groups) who underwent lumbar disc surgery between 25 july 2022-30 december, 2022. Data will be collected with Introductory Information Form, Visual Comparison Scale, Oswestry Disability Index, Functional Low Back Pain Scale, Medication Tracking Form, Tape Tracking Form, Gait Tracking Form, "Healing Process After Lumbar Hernia Surgery".

The taping process will be done by the researcher Gülşah Bilgin, who has attended the course after receiving training on this subject.

All participants in the study will be informed about the study on the first day of their hospitalization, and the Introductory Information Form, Visual Comparison Scale, and Oswestry Disability Index will be filled by the patients, and the researcher will assist the patients who are illiterate or have difficulty in understanding the questions. 24 hours after the operation, a brochure will be given to the patients and their relatives, included in the study by the sampling inclusion and exclusion criteria, to provide a 20-minute education and reminder about the use of a pedometer and home care during the rehabilitation process after herniated disc surgery. Visual Analogue Scale, Oswestry Disability Index, and Functional Low Back Pain Scale for the first follow-up will be filled and all medications taken by the patient, including analgesics, will be recorded on the Medication Tracking Form.

During the treatment and follow-up periods, the use of drugs will not be restricted and they will be asked to record the drugs used. The individuals participating in the study will not be informed about which group they belong to. After the Kinesio/placebo tape application, the patients and their relatives will be shown how to fill out the Medication Follow-up Form and the Walking Follow-up Form.

It is designed by the nurse to facilitate the natural healing process after trauma/inflammation by providing stability and support to the muscles and joints in patients who may experience moderate pain, disability and loss of functionality after lumbar disc surgery.

The aim of this study was to examine the efficacy and safety of the kinesio tape to be applied in reducing pain and maintaining functionality.

Tape will be applied to the placebo and kinesio groups four times and for five days each time. In both groups, the application days and durations of the kinesio tape will be the same, only the application method of the tape will differ. The application will be made in the surgical clinic of a public hospital. exercise to work Patients who do not have a disability, who do not have chronic diseases such as neurological problems, respiratory heart failure, diabetes, and who have undergone standard discectomy will participate. Patients who underwent standard discectomy in the first 24 hours post-op were randomized to one of the two groups.

will be made. In the study, band application will be performed 4 times in 30 days and pain and functionality assessment will be made.

Evaluation of the data: Evaluation of the data will be done in the computer environment, and parametric and nonparametric tests will be used according to the number, percentage, mean, median, and normality distribution from introductory statistics. p ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-65,
* Having had standard discectomy surgery in the last 24 hours, and
* To sign the Informed Voluntary Consent Form.

Exclusion Criteria:

* Having had surgery other than standard laminectomy or discectomy surgery in the last 24 hours,
* Complications developed in the early postoperative period (such as severe bleeding, nausea, vomiting, hemiplegia),
* Having undergone spinal surgery before,
* To have applied Kinesio tape treatment,
* To have received corticosteroid treatment in the two weeks before the surgery, Having clinical signs of central or peripheral nervous system disease (such as sensitivity to touch, lack of coordination, pain even in normal activities, memory loss),
* Being pregnant, Being under the age of 18 and over the age of 65,
* Having a neurological or orthopedic problem that may adversely affect the evaluation of exercise capacity, Having been diagnosed with respiratory or heart failure, and Having insulin-dependent diabetes and
* Not signing the Informed Consent Form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the 10-point Visual Analog Scale at Day 30. | Baseline and Day 1, 5, 10, 15, 30.
  The visual analogue scale is a 10cm ruler that shows "painlessness" at one end and "the most severe pain possible" at the other end. Change= (day 30- Baseline score)
pain - Medication tracking form | from the postoperative period to the 30th day
  All drugs used by the patient will be recorded on the drug form by the researcher at the hospital and by the patient or their relatives after they go home.The average score for painkillers will be evaluated as 2 points for narcotics and 1 point for non-narcotic drugs. The score will be calculated according to the dose taken by the patient, and if the patient has taken narcotic analgesics 2 times a day, the score will be 4 points.An increase in the score will be interpreted as an increase in the level of pain.

SECONDARY OUTCOMES:
functionality-Oswestry Disability Index at Day 30. | Baseline and Day 5, 10, 15, 30.
  The Oswestry Disability Index is an outcome-based self-assessment scale developed to assess low back pain. According to this index, "0" is the lowest score and "50" is the highest score. The total score is multiplied by two and expressed as a percentage. If the average score to be obtained from the scale is between 0-10 points, it is accepted as "low level disability", and between 11-30 points as "moderate disability". , and 31-50 points "severe injury". A 6-point improvement on the Oswestry scale is considered a "significant effect" in individuals with low back pain.
functionality-Functional Low Back Pain Scale | Day 1, 5, 10, 15, 30.
  The Functional Low Back Pain Scale is a scale that aims to evaluate the functional status and daily activities of the person, changes in functional status such as bending forward, sitting, standing, walking, climbing stairs and driving.is being done.Each item is scored between 0 and 5; Scoring is "0" not possible to do the activity, "5 points" not difficult. The possible score ranges from 0 to 60. The increase in the score shows that the performance activity is not difficult.
functionality-Pedometer | Day 5, 10, 15, 30.
  Pedometer is a device used to evaluate physical activity performance.The average number of steps per day; The average was calculated by dividing the total number of daily steps between day 1 and day 5 by four.
Evaluation of healing at the surgical site-Kinesio follow-up form | Day 1, 5, 10, 15, 30.
  In the evaluation of wound healing, the condition of the wound edges according to the days (epithelialization 1 point, open 0 points), bleeding (hemorrhage 1 point not 0 points), tenderness (tenderness 1 point, no 0 points), infection (1 point not present, 0 points) ), color (normal skin color 1 point, redness 01 points, purulent 02 points), edema (1 point, no 0 points), ecchymosis (1 point, no 0 points), fever (1 point, no 0 points). evaluated over. In the evaluation of the side effects of the kinesio tape, it was evaluated according to skin reactions (1 point, 0 point not present), allergic reaction status (1 point, 0 point not present).An increase in the score compared to the baseline will be interpreted as worsening wound healing, while a decrease will be interpreted as improving wound healing.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Öncü, pHD, Principal Investigator — Mersin University; Melih Çekinmez, pHD, Principal Investigator — Adana Şehir Hastanesi
Locations (1):
- SBÜ Adana Şehir Eğitim ve Araştırma Hastanesi, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bilgin G, Oncu E, Cekinmez M. The Effect of I-Shaped Kinesiotaping on Pain, Functionality, and Wound Healing After Lumbar Disc Surgery: A Randomised Controlled Trial. Biol Res Nurs. 2026 Jan 13:10998004261416820. doi: 10.1177/10998004261416820. Online ahead of print. PMID 41528353